CLINICAL TRIAL: NCT06057701
Title: Effect of Exercises on Diaphragmatic Excursion in Postmenopausal Kyphotic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samia Samir Rashed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: postmenopausal kyphosis
Record Dates: First submitted 2023-09-17; First posted 2023-09-28 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Kyphosis Postural Thoracic
Keywords: postmenopausal kyphosis; flexicurve ruler; diaphragmatic excursion; corrective exercises; resisted diaphragmatic breathing

STUDY DESIGN:
Intervention Model Description: intervention:
  Group A:
  This group was consisted of 20 postmenopausal women suffering from thoracic kyphosis. They received corrective exercises for twice a week for 12 weeks.
  corrective exercises: The patient did a daily session of 20-30 min (under the supervision of the therapist or alone at home). It consisted of warm up phase for 5 minutes (breathing exercises), active phase (corrective exercises) and cooling down phase finally for return to the initial state.
  strengthening exercises and stretching exercise
  Group B:
  The study group consisted of 20 postmenopausal women suffering from thoracic kyphosis, who received corrective exercises prescribed above in addition to resisted diaphragmatic breathing exercise.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): This group consists of 20 postmenopausal women suffering from thoracic hyper kyphosis. They receive daily session of 30minutes even by therapist or at home for 12 weeks. the corrective exercises for the thoracic spine consist of strengthening exercises for back muscles and stretching exercises for pectoral muscles
  Interventions: Other: corrective exercises
- interventional group (Experimental): This group consists of 20 postmenopausal women suffering from thoracic hyper kyphosis, who receive the corrective exercises prescribed above in addition to resisted diaphragmatic breathing exercise. They receive daily session of 30minutes even by therapist or at home for 12 weeks.
  Interventions: Other: corrective exercises; Other: resisted diaphragmatic breathing exercises

INTERVENTIONS:
Other: corrective exercises — corrective exercises:
  1. Strengthening exercises :
     1. Thoracic extension exercises:
        * Mckanzie's thoracic extension exercise:
        * Thoracic spine stretching position
     2. Back extension exercise
     3. Abdominal curl up exercise
     4. Scapular retraction exercises
     5. Trunk rotation exercise
  2. Stretching exercises:
     1. Pectoral muscles stretch from sitting
     2. self-stretch for pectoral muscle infront of door
Other: resisted diaphragmatic breathing exercises — 1. Diaphragmatic breathing exercise: From the supine position, overlapping hands on the diaphragm located in the abdominal region: each woman took deep inspiring by the nose and exhaling through the mouth with lips half-closed slowly.
  2. Resisted diaphragmatic breathing exercise: From the supine position, with a weight of 1 kg on the diaphragm located in the abdominal region: each woman took deep inspiring by the nose and exhaling through the mouth with lips half-closed slowly
  Arms: interventional group

SUMMARY:
the present study examined the effect of different types of exercises for improving the age-related hyperkyphotic curve of postmenopausal women and also examined how it affects diaphragmatic excursion and respiratory function. Increasing the respiratory functions for elderly will act as a preventive method against nowadays chest diseases.

DETAILED DESCRIPTION:
The study was conducted to examine the effect of exercises on diaphragmatic excursion in postmenopausal kyphotic women.

Design of study:

A prospective, randomized, single-blind, pre-post-test, controlled trial. The study followed the Guidelines of Declaration of Helsinki on the conduct of human research. Ethical approval was obtained from the institutional review board at Faculty of physical therapy, Cairo University before study commencement (no.P.T,REC/012/003800).

This study was carried on forty postmenopausal women clinically diagnosed with thoracic kyphosis. They selected randomly from the outpatient clinic of El Kaser El-Einy University Hospital, Cairo University. Their ages ranged from 50-60 years.

Randomization of sample selection was achieved using closed envelop way. Classification of the sample by simple random way into two groups equal in number, twenty for each group by using forty closed envelop, each twenty envelop contained a name of a group from the two groups (Group A) or (Group B) and asking each woman to choose one envelop from them, each woman attended to the group according the name of the group written in her envelop.

ELIGIBILITY:
Inclusion Criteria:

1. All postmenopausal women suffering from thoracic kyphosis.
2. Their thoracic kyphosis (Cobb's) angles were more than 45 degrees.
3. Their age ranged from 50-60 years old.
4. Their BMI were >25 and <30 kg/m2.

Exclusion Criteria:

1. All patients with comorbidities such as cardiac disease and chest diseases as pulmonary fibrosis.
2. Patients with previous trauma to the spine, pelvis and lower limbs.
3. Patients with a previous history of spinal surgery (such as spinal fusion surgery, vertebroplasty, or kyphoplasty).
4. Patients with congenital spinal deformities and scoliosis.
5. Patients with a history of spinal tumors, ankylosing spondylitis, osteoporosis and other spondyloarthritis.
6. The patients received medications that might affect the neuromuscular functions at least three months before or during the study course.
7. Patients suffered from mental or psychological disorders.
8. Patients suffered from inflammatory diseases such as rheumatoid arthritis or polymyalgia rheumatic.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
flexicurve ruler | period of treatment is for 12 weeks
  A flexible curve ruler was used to measure the kyphosis angle. The adjustable curve is one of the non-invasive methods for kyphosis and lordosis angle assessments in the sagittal plan.
Diaphragmatic excursion | period of treatment is for 12 weeks
  To measure diaphragmatic excursion, an ultrasonography device was applied with a probe frequency of 2-5 MHz. The right hemi-diaphragmatic excursion was assessed during deep inspiration and deep expiration
Quality of life questionnaire of the European foundation for osteoporosis (QUALEFFO-41) | period of treatment is for 12 weeks
  The QUALEFFO-41 is a self-administered, disease specific questionnaire used frequently in clinical research. It possesses five domains (41 items in total): pain (5 items), physical function (17 items), social function (7 items), general health perception (3 items) and mental function (9 items).
  The total QUALEFFO score is calculated as a sum of all answers to items and then linearly transformed on the scale 0-100. The worse the HRQOL condition is, the higher the score gets. The actual score was calculated by the summation of all questions answers, the lowest possible score was 41, the score range was 164 (41 subtracted from 205)
Pain assessment scale | period of treatment is for 12 weeks
  Visual analogue scale (VAS) is the most common pain scale for quantification of endometriosis-related pain and skin graft donor site-related pain. A review came to the conclusion that VAS was one of the best adapted pain scales for pain measurement for research purposes.The scale described by the researcher to patients in order to make its use easy. The patients will chose a value from numerized values from 0-10 printed on the scale, 0 (indicates no pain) while 10 (indicates maximum pain) and in between the values are classified.

CONTACTS AND LOCATIONS:
Overall Officials: Fahima okeel, Study Chair — Cairo University; Amal Yousef, Study Director — Cairo University; Khaled Kamel, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt